CLINICAL TRIAL: NCT03132545
Title: Resting Metabolic Rate, Fat Distribution, Endocrine and Metabolic Features in Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Valeria Tagliaferri, Dr, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ARMOC
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS
  Interventions: Diagnostic Test: SenseWear Armband (SWA) monitoring; Diagnostic Test: total body dual-energy X-ray absorptiometry
- controls
  Interventions: Diagnostic Test: SenseWear Armband (SWA) monitoring; Diagnostic Test: total body dual-energy X-ray absorptiometry

INTERVENTIONS:
Diagnostic Test: SenseWear Armband (SWA) monitoring — Participants wore the SWA on their right arm
Diagnostic Test: total body dual-energy X-ray absorptiometry — DEXA was used to estimate abdominal visceral adipose tissue and subcutaneous adipose tissue

SUMMARY:
In a longitudinal, prospective and observational study, patients with PCOS and controls wore the SenseWear Armband for 2 days. Resting metabolic rati (kcal/die), total energy expenditure (MET, kcal) were evaluated. Ultrasonographic pelvic examinations, hirsutism score, anthropometric and menstrual pattern evaluation, hormonal profile assays, oral glucose tolerance test (OGTT) and lipid profile were performed.

ELIGIBILITY:
Inclusion Criteria:

* . PCOS diagnosed according with the Rotterdam Consensus Conference criteria

Exclusion Criteria:

* presence of a late-onset adrenal enzyme defect
* Significant liver or renal impairment
* pregnancy and nursing
* neoplasm
* cardiovascular disease
* other hormonal dysfunctions

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: group 1: women with PCOS diagnosed according with the Rotterdam Consensus Conference criteria group 2: healty women
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
differences in resting metabolic rate | 2 days

SECONDARY OUTCOMES:
differences in body fat distribution | 1 day

REFERENCES:
- [Derived] Romualdi D, Versace V, Tagliaferri V, De Cicco S, Immediata V, Apa R, Guido M, Lanzone A. The resting metabolic rate in women with polycystic ovary syndrome and its relation to the hormonal milieu, insulin metabolism, and body fat distribution: a cohort study. J Endocrinol Invest. 2019 Sep;42(9):1089-1097. doi: 10.1007/s40618-019-01029-2. Epub 2019 Mar 7. PMID 30847861